CLINICAL TRIAL: NCT02362997
Title: A Phase 2 Study of Pembrolizumab (MK-3475) After Autologous Stem Cell Transplantation in Patients With Relapsed/Refractory Classical Hodgkin Lymphoma and, Diffuse Large B Cell Lymphoma and T- Cell Non-Hodgkin Lymphoma
Brief Title: Pembrolizumab After ASCT for Hodgkin Lymphoma, DLBCL and T-NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-566
Record Dates: First submitted 2015-02-05; First posted 2015-02-13 (Estimated); Results first posted 2022-12-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2023-07

CONDITIONS: Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Peripheral T-Cell Lymphoma
Keywords: Classical Hodgkin Lymphoma (cHL); Diffuse Large B Cell Lymphoma (DLBCL); Peripheral T-cell lymphoma (PTCL)
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diffuse large B cell lymphoma (Experimental): Pembrolizumab 200mg IV every 3 weeks up to 8 cycles
  Interventions: Drug: Pembrolizumab
- Classical Hodgkin lymphoma (Experimental): Pembrolizumab 200mg IV every 3 weeks up to 8 cycles
  Interventions: Drug: Pembrolizumab
- Peripheral T cell lymphoma (Experimental): Pembrolizumab 200mg IV every 3 weeks up to 8 cycles
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Anti-PD-1 monoclonal antibody
  Other Names: Keytruda; MK-3475; SCH 900475

SUMMARY:
This phase II study is designed to determine the clinical efficacy of PD-1 blockade, using the anti-PD-1 monoclonal antibody pembrolizumab (MK-3475), administered as consolidation therapy after autologous stem cell transplant (ASCT), in patients with relapsed or refractory (R/R) Diffuse Large B Cell Lymphoma (DLBCL), classical Hodgkin Lymphoma (cHL) or peripheral T-cell lymphoma (PTCL) in 1st remission.

DETAILED DESCRIPTION:
Pembrolizumab is an antibody drug that blocks a molecule called PD-1. PD-1 is a receptor molecule on the surface of immune cells that can be used to turn off the immune response. Some cancers use this as a way to turn off the immune response against them. Blocking PD-1 with pembrolizumabmay restore an effective immune attack against the lymphoma cells.

On this study, patients who undergo ASCT for R/R cHL, DLBCL or PTCL in 1st remission will receive pembrolizumab at a dose of 200mg intravenously every 3 weeks for up to 8 cycles, beginning within a few weeks of ASCT.

ELIGIBILITY:
Inclusion criteria

• Histologically confirmed diagnosis with review of the diagnostic pathology specimen at one of the participating institutions. Eligible histologies are: Arm A: Diffuse large B cell lymphoma; patients with a prior history of indolent B-cell NHL are eligible, as long as they have histologically confirmed DLBCL prior to their pre-transplant salvage treatment. Patients with mediastinal large B cell lymphoma are also eligible.

Arm B: Classical Hodgkin lymphoma (patients with nodular lymphocyte predominant Hodgkin lymphoma [NLPHL] are NOT eligible) Arm C: Peripheral T cell lymphoma - eligible subtypes will include PTCL, NOS; AITL; and ALK-negative ALCL. Patients with other PTCL histologies, including ALK-positive PTCL, and cutaneous T-cell lymphoma will not be eligible..

* Age ≥ 18 at the time of enrollment.
* For arms A and B, participants must have relapsed after or been refractory to first-line chemotherapy, i.e., they must have failed to achieve CR after first-line therapy or must have relapsed subsequently if they achieved CR. For arm C, participants will be eligible if transplant is performed as consolidation of first remission (partial or complete).
* Participants must be planning to receive or have received autologous stem cell transplantation. Participants must have chemosensitive disease prior to ASCT, defined as achieving at least a partial remission (as determined with PET imaging) to salvage treatment. Participants with cHL or DLBCL (arms A and B) transplanted in 1st remission after only one line of treatment are not eligible. Participants with PTCL (arm C) transplanted beyond 1st remission are also not eligible.
* No more than 1 line of anthracycline-containing chemotherapy prior to ASCT, and no more than 3 lines of therapy total prior to ASCT for arms A and B; no more than 1 line of therapy prior to ASCT for arm C.
* Participants cannot have received any anti-neoplastic therapy (including radiotherapy, chemotherapy or immunotherapy) after ASCT
* Participants must have had PET-CT for restaging after salvage therapy and before ASCT.
* Participants must begin study treatment no later than 21 days from the post-ASCT discharge. Additionally, they must have recovered from ASCT toxicities at the time of first study treatment.
* ECOG performance status ≤2
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 50,000/mcL
  * Hemoglobin ≥ 8 g/dl
  * total bilirubin ≤ 1.5 × institutional upper limit of normal (ULN), or direct bilirubin ≤ ULN in patients with Gilbert's syndrome
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × ULN
  * Creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 60 mL/min/1.73 m2
  * Resting and ambulatory oxygen saturation ≥ 94% on room air
  * FEV1 and DLCO (adjusted for Hemoglobin) ≥ 50% predicted
* Willigness to use contraception
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion criteria

* Participants who are receiving any other investigational agents after ASCT.
* Participants with active CNS involvement are excluded.
* History of or active autoimmune disease, or other syndrome that requires systemic steroids or autoimmune agents. Participants with vitiligo, resolved childhood asthma or atopy, hypothyroidism, or Sjogren's syndrome, as well as participants requiring only intranasal steroids, intermittent use of bronchodilators, local steroid injections, or physiologic replacement doses of prednisone (≤ 10 mg/d) are not excluded from this study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab. Prior hypersensitivity reactions to anti-CD20 therapy or anti-CD30 therapy is not an exclusion criterion.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Receipt of > 600 mg/m2 total dose of BCNU with prior treatments including transplant conditioning regimen.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements or pose excess risk to the participant in the opinion of the treating clinician..
* Pregnant or lactating women.
* HIV-positive.
* Participants with active viral hepatitis (positive HepB sAg, positive HepB core Ab with positive HepB viral load, or positive HepC antibody with positive HepC viral load).
* Receipt of a live vaccine within 30 days of the start of treatment. Examples are measles, mumps, rubella, varicella, yellow fever, rabies, BCG, oral polio vaccine, and oral typhoid vaccine.
* Prior treatment with an anti PD-1, anti PD-L1, or anti CTLA-4 agent. Participants who entered clinical remission with one of those agents and proceeded to ASCT without intervening relapse may be eligible after discussion with the Study Chair. Note that for patients who enter remission with checkpoint blockade therapy, this will not count towards the 3 lines of prior therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-04; Primary Completion 2021-10-26 (Actual); Study Completion 2023-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Armand, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - City of Hope National Medical Center, Duarte, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Merrill MH, Dahi PB, Redd RA, McDonough MM, Chen YB, DeFilipp Z, Herrera AF, Fisher DC, LaCasce AS, Odejide OO, Ng SY, Jacobson CA, Merryman RW, Kim AI, Nieto YL, Sauter CS, Shah GL, Zain JM, Armand P, Jacobsen ED. A phase 2 study of pembrolizumab after autologous stem cell transplantation in patients with T-cell non-Hodgkin lymphoma. Blood. 2023 Aug 17;142(7):621-628. doi: 10.1182/blood.2023020244. PMID 37319432
- [Derived] Merryman RW, Redd RA, Taranto E, Ahmed G, Jeter E, McHugh KM, Brown JR, Crombie JL, Davids MS, Fisher DC, Freedman AS, Jacobsen E, Jacobson CA, Kim AI, LaCasce AS, Ng SY, Odejide OO, Parry EM, Jacene H, Park H, Dahi PB, Nieto Y, Joyce RM, Chen YB, Shipp MA, Herrera AF, Armand P. Minimal residual disease in patients with diffuse large B-cell lymphoma undergoing autologous stem cell transplantation. Blood Adv. 2023 Sep 12;7(17):4748-4759. doi: 10.1182/bloodadvances.2022007706. PMID 36399518
- [Derived] Merryman RW, Redd R, Jeter E, Wong JL, McHugh K, Reynolds C, Nazzaro M, Varden A, Brown JR, Crombie JL, Davids MS, Fisher DC, Jacobsen E, Jacobson CA, Kim AI, LaCasce AS, Ng SY, Odejide OO, Parry EM, Dahi PB, Nieto Y, Joyce RM, Chen YB, Herrera AF, Armand P, Ritz J. Immune Reconstitution following High-Dose Chemotherapy and Autologous Stem Cell Transplantation with or without Pembrolizumab Maintenance Therapy in Patients with Lymphoma. Transplant Cell Ther. 2022 Jan;28(1):32.e1-32.e10. doi: 10.1016/j.jtct.2021.10.010. Epub 2021 Oct 17. PMID 34670169
- [Derived] Frigault MJ, Armand P, Redd RA, Jeter E, Merryman RW, Coleman KC, Herrera AF, Dahi P, Nieto Y, LaCasce AS, Fisher DC, Ng SY, Odejide OO, Freedman AS, Kim AI, Crombie JL, Jacobson CA, Jacobsen ED, Wong JL, Bsat J, Patel SS, Ritz J, Rodig SJ, Shipp MA, Chen YB, Joyce RM. PD-1 blockade for diffuse large B-cell lymphoma after autologous stem cell transplantation. Blood Adv. 2020 Jan 14;4(1):122-126. doi: 10.1182/bloodadvances.2019000784. PMID 31917843
- [Derived] Armand P, Chen YB, Redd RA, Joyce RM, Bsat J, Jeter E, Merryman RW, Coleman KC, Dahi PB, Nieto Y, LaCasce AS, Fisher DC, Ng SY, Odejide OO, Freedman AS, Kim AI, Crombie JL, Jacobson CA, Jacobsen ED, Wong JL, Patel SS, Ritz J, Rodig SJ, Shipp MA, Herrera AF. PD-1 blockade with pembrolizumab for classical Hodgkin lymphoma after autologous stem cell transplantation. Blood. 2019 Jul 4;134(1):22-29. doi: 10.1182/blood.2019000215. Epub 2019 Apr 5. PMID 30952672

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Started | 31 | 30 | 21
Completed | 31 | 30 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma | Total
Number analyzed (Participants) | 31 | 30 | 21 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 29 | 15 | 67
  >=65 years | 8 | 1 | 6 | 15
Age, Continuous [Median (Full Range); unit: years] | 57 [22 to 76] | 34 [20 to 69] | 58 [33 to 73] | 50 [20 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 9 | 32
  Male | 22 | 16 | 12 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 24 | 18 | 13 | 55
  Unknown or Not Reported | 6 | 12 | 8 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 25 | 17 | 10 | 52
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 4 | 12 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 21 | 82
ECOG Performance Score [Count of Participants; unit: Participants]
  00- Fully Active | 10 | 14 | 4 | 28
  01- Restricted | 20 | 16 | 16 | 52
  02- Ambulatory and Capable of Self Care | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival After ASCT
Description: Proportion of patients alive and disease-free 18 months from autologous stem cell transplantation (ASCT). Progression criteria are per Lugano 2014 criteria. All patients receiving any amount of protocol treatment. Patients who have progressed or lost to follow-up prior to 18 months are counted as failures; only patients followed and progression-free for at least 18 months are counted as successes.
Time Frame: 18 Months
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 31 | 30 | 21
proportion of participants | 0.58 [0.42 to 0.73] | 0.77 [0.61 to 0.89] | 0.62 [0.42 to 0.79]

2. Secondary Outcome: Overall Survival
Description: Survival probability of patients alive 18 months from ASCT, time-to-event
Time Frame: 18 Months
Measure: Number (90% Confidence Interval); unit: survival probability
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 31 | 30 | 21
survival probability | 0.93 [0.85 to 1.0] | 1.0 [1.0 to 1.0] | 0.94 [0.86 to 1.0]

3. Secondary Outcome: Relapse
Description: Number of patients who relapse within 18 months from autologous stem cell transplantation.
Time Frame: 18 Months
Population: Patients who have been followed for at least 18 months or have relapsed prior to 18 months post ASCT
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 25 | 28 | 16
Participants | 11 | 4 | 4

4. Secondary Outcome: Safety and Tolerability Assessed by CTCAE v4 Grade 2 and Above Toxicity Related to Study Treatment
Description: Number of patients who experienced at least a grade 2 toxicity with "definite," "probable," or "possible" attribute to study treatment, according to the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 31 | 30 | 21
Participants | 21 | 15 | 12

5. Secondary Outcome: Response Rate to Pembrolizumab
Description: In patients with measurable disease after ASCT, rate of objective response after treatment. Response was assessed using the Lugano 2014 criteria.
Time Frame: 18 months
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 31 | 30 | 21
proportion of participants | 0.74 [0.58 to 0.86] | 0.90 [0.76 to 0.97] | 0.86 [0.67 to 0.96]

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival probability of patients who are alive and without progression 18 months from ASCT, time-to-event
Time Frame: 18 months
Measure: Number (90% Confidence Interval); unit: progression-free survival probability
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 31 | 30 | 21
progression-free survival probability | 0.74 [0.62 to 0.90] | 0.87 [0.77 to 0.97] | 0.84 [0.70 to 0.99]

7. Other Pre Specified Outcome: Overall Survival After ASCT by PET Status
Description: Survival probability of patients alive 18 months from ASCT stratified by PET status before transplantation, time-to-event. Patients categorized by complete metabolic response (complete response by PET scan, assessed using the Lugano 2014 criteria), partial response (assessed using Lugano 2014 criteria) prior to transplantation.
Time Frame: 18 months
Measure: Number (90% Confidence Interval); unit: survival probability
Groups:
- Diffuse Large B Cell Lymphoma, PET-CR: Diffuse Large B Cell Lymphoma patients who were PET-CR before transplantation
- Diffuse Large B Cell Lymphoma, PET-NCR: Diffuse Large B Cell Lymphoma patients who were not PET-CR before transplantation
- Classical Hodgkin Lymphoma - PET-CR: Classical Hodgkin Lymphoma patients who were PET-CR before transplantation
- Classical Hodgkin Lymphoma - PET-NCR: Classical Hodgkin Lymphoma patients who were not PET-CR before transplantation
- Peripheral T Cell - PET-CR: Peripheral T Cell patients who were PET-CR before transplantation
- Peripheral T Cell - PET-NCR: Peripheral T Cell patients who were not PET-CR before transplantation
Arm/Group | Diffuse Large B Cell Lymphoma, PET-CR | Diffuse Large B Cell Lymphoma, PET-NCR | Classical Hodgkin Lymphoma - PET-CR | Classical Hodgkin Lymphoma - PET-NCR | Peripheral T Cell - PET-CR | Peripheral T Cell - PET-NCR
Number analyzed (Participants) | 20 | 11 | 23 | 7 | 19 | 2
survival probability | 0.94 [0.85 to 1.0] | 0.91 [0.78 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 0.94 [0.84 to 1.0] | 1.0 [1.0 to 1.0]

8. Other Pre Specified Outcome: Progression-free Survival After ASCT by PET Status
Description: Progression-free survival probability of patients alive and disease-free 18 months from ASCT stratified by PET status before transplantation, time-to-event
Time Frame: 18 months
Measure: Number (90% Confidence Interval); unit: progression-free survival probability
Arm/Group | Diffuse Large B Cell Lymphoma, PET-CR | Diffuse Large B Cell Lymphoma, PET-NCR | Classical Hodgkin Lymphoma - PET-CR | Classical Hodgkin Lymphoma - PET-NCR | Peripheral T Cell - PET-CR | Peripheral T Cell - PET-NCR
Number analyzed (Participants) | 20 | 11 | 23 | 7 | 19 | 2
progression-free survival probability | 0.87 [0.74 to 1.0] | 0.54 [0.35 to 0.86] | 0.82 [0.70 to 0.97] | 1.0 [1.0 to 1.0] | 0.82 [0.67 to 0.99] | 1.0 [1.0 to 1.0]

9. Other Pre Specified Outcome: Completion Rate
Description: Number of patients who complete the planned treatment
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
Number analyzed (Participants) | 31 | 30 | 21
Participants | 18 | 23 | 14

10. Other Pre Specified Outcome: Minimal Residual Disease
Description: Level of MRD detected by PCR (if feasible) before and after pembrolizumab
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Safety assessments will be performed on day 1 of each of up to 8 treatment cycles (28-day cycle) followed by assessments every 3 months until up to 18-months post-ASCT
Arm/Group | Diffuse Large B Cell Lymphoma | Classical Hodgkin Lymphoma | Peripheral T Cell Lymphoma
All-Cause Mortality (participants affected / at risk) | 2/31 | 0/30 | 3/21
Serious Adverse Events (participants affected / at risk) | 8/31 | 3/30 | 1/21
Other Adverse Events (participants affected / at risk) | 29/31 | 30/30 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diffuse Large B Cell Lymphoma (N=31) | Classical Hodgkin Lymphoma (N=30) | Peripheral T Cell Lymphoma (N=21)
Neutrophil count decreased (Investigations) | 6 (6) | 3 (4) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Right neck mass
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Squamous cell carcinoma
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Airway compromise
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diffuse Large B Cell Lymphoma (N=31) | Classical Hodgkin Lymphoma (N=30) | Peripheral T Cell Lymphoma (N=21)
Fatigue (General disorders) | 17 (24) | 15 (17) | 13 (18)
Anemia (Blood and lymphatic system disorders) | 18 (32) | 14 (29) | 11 (22)
Platelet count decreased (Investigations) | 19 (37) | 9 (18) | 7 (13)
Diarrhea (Gastrointestinal disorders) | 14 (23) | 7 (11) | 11 (18)
Nausea (Gastrointestinal disorders) | 12 (19) | 8 (12) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 11 (13) | 6 (7)
Neutrophil count decreased (Investigations) | 15 (25) | 7 (9) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (19) | 7 (7) | 4 (4)
Alanine aminotransferase increased (Investigations) | 10 (12) | 9 (23) | 3 (10)
Aspartate aminotransferase increased (Investigations) | 10 (11) | 8 (13) | 3 (8)
White blood cell decreased (Investigations) | 9 (19) | 9 (24) | 2 (6)
Upper respiratory infection (Infections and infestations) | 9 (15) | 10 (14) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 5 (7) | 6 (11)
Alkaline phosphatase increased (Investigations) | 5 (8) | 5 (8) | 5 (10)
Dizziness (Nervous system disorders) | 5 (8) | 4 (7) | 6 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (6) | 7 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (12) | 3 (3) | 3 (3)
Fever (General disorders) | 6 (6) | 6 (7) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 3 (3) | 6 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6) | 4 (5) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 6 (9)
Constipation (Gastrointestinal disorders) | 4 (4) | 2 (2) | 6 (6)
Hypertension (Vascular disorders) | 9 (17) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 5 (6) | 2 (2)
Hypothyroidism (Endocrine disorders) | 2 (2) | 4 (8) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 6 (12)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6) | 5 (8) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5) | 5 (7) | 1 (1)
Pain (General disorders) | 4 (4) | 4 (5) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (5) | 4 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (6)
Dysgeusia (Nervous system disorders) | 3 (4) | 0 (0) | 5 (6)
Chills (General disorders) | 4 (4) | 2 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (4) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 5 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (2) | 2 (4)
Lung infection (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 5 (9) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 2 (4)
Paresthesia (Nervous system disorders) | 2 (4) | 0 (0) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (3)
Weight loss (Investigations) | 1 (2) | 0 (0) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 3 (3)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1) — Itchy jawbone and cheeks, Psoriasis, Red facial nodule secondary to spa treatment, Bump on scalp, Rash
Edema limbs (General disorders) | 1 (3) | 0 (0) | 3 (4)
Colitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) — Herpes Zoster left leg pain, Influenza infection, Influenza Type A, COVID-19
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02362997/Prot_SAP_000.pdf